CLINICAL TRIAL: NCT03041103
Title: Acceptability and Tolerance of a Protein and Micronutrient Fortified Nutritious Food Product in Californian Adults and Children
Brief Title: Acceptability and Tolerance of a Protein and Micronutrient Fortified Food
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 985880
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Poor Nutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Single arm not blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult (Experimental): Food Product 1:50 grams of fortified nutritious product from legumes administered to adults, for 2 weeks
  Interventions: Other: Food Product 1
- Children (Experimental): Food Product 1: 50 grams of fortified nutritious product from legumes administered to children 9-13 years of age, for 1 weeks
  Interventions: Other: Food Product 1

INTERVENTIONS:
Other: Food Product 1 — 50 grams of fortified nutritious product from legumes

SUMMARY:
Acceptability and tolerance of a new food product in adults and children.

DETAILED DESCRIPTION:
Acceptability and tolerance testing will be conducted in 10 healthy male adult volunteers and 10 (40 - 60 years of age), and in children (9-13 years of age). All participants will be asked to consume 50g of a test product every day for 2 weeks for the adult volunteers, while the children will be asked to consume the same product every day for one week. The participants will record amount of daily intake, and will be given an entry and exit surveys. These surveys will include the assessment of potential gastrointestinal changes with daily product intake, and will include questions on how they liked the product. Acceptability will be measured as the number of servings and portion of serving completed each day over the trial period.

In adults only, fasting blood samples and a spot urine will be collected towards preliminary work on potential changes in the metabolome and lipidome with the inclusion of the test product within the habitual diet.

ELIGIBILITY:
° Inclusion Criteria:

* Male, 40-60 years old
* Male or Female 9-13 years old
* Subject is willing and able to comply with the study protocols
* Subject is willing to consume the test products

Exclusion Criteria:

* Allergies or intolerances to peas, legumes, pulses, soy, dairy or wheat/gluten
* Under current medical supervision
* Non-English speaking
* Self-reported history of cardiovascular disease, stroke, cancer, renal, hepatic, or thyroid disease, GI tract disorders, previous GI surgery
* Currently taking prescription drugs or supplements
* Daily use of aspirin and or non-steroidal anti-inflammatory medicines.
* Indications of substance or alcohol abuse within the last 3 years
* Any supplement use, including multi-vitamin/ mineral, herbal, plant or botanical, fish oil, and oil supplements.
* Self-reported malabsorption
* Current enrollee in a clinical research study.

Ages: 9 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
GI function | at 2 weeks
  GI function questionnaire with categorical numerical score

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Department of Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No